CLINICAL TRIAL: NCT06537453
Title: Using Personalized Risk and Digital Tools to Guide Transitions Following Acute Kidney Events - Virtual Care: Virtual Home Hospital With Remote Monitoring to Reduce Acute Care Hospitalization
Brief Title: UPTAKE - Virtual Care: Virtual Home Hospital With Remote Monitoring to Reduce Acute Care Hospitalization
Acronym: UPTAKE-VC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REB23-0762
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: One group will receive the Virtual Care Intervention through Virtual Home Hospitals and other group will receive Usual Care.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized in either arm, will be coded such that the outcome assessor is blinded to the arm assignment of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Care (Experimental): Participants will receive virtual care through Virtual Home Hospital programs in Alberta for their hospital to home transition of care.
  Interventions: Other: Virtual Care
- Usual Care (No Intervention): Participants will be discharged as per usual care practices from hospital to their home.

INTERVENTIONS:
Other: Virtual Care — Participants will go through Virtual hospital programs following the processes established by these programs in Alberta.
  Arms: Virtual Care

SUMMARY:
Method: Randomized Controlled Trial Study Duration: 3 Years Study Centre(s) University of Calgary and University of Alberta Objectives: To fill care gaps by implementing strategies to reduce length of hospital stay, readmission rates, and improve long-term outcomes after Acute Kidney Injury (AKI). Number of Participants: Three Hundred and fifty four (n=354) Diagnosis and Main Inclusion Criteria: Hospitalized adults with AKI at high risk of hospital readmission or death

Study Intervention: Multi-component Digital Health Solutions, including:

1. Computerized Clinical Decision Support (CDS) and
2. Virtual Care Delivered through Hospital at Home (VC) Duration of administration: Determined by the Patient's clinical team Reference therapy: Usual Care Statistical Analyses: Descriptive Analysis, Regression

DETAILED DESCRIPTION:
1. Background and Rationale

   Acute kidney injury (AKI) is a common and serious complication in hospitals. A major care gap for survivors of AKI is the fragmentation of care that exists as they transition from the hospital to their home. This contributes to a high risk of adverse long-term outcomes, including prolonged hospitalization, high rates of readmission, cardiovascular events, infections, progression to chronic kidney disease (CKD), kidney failure requiring dialysis, and death.

   To address this challenge, the investigators are implementing multi-component digital health solutions including Computerized Clinical Decision Support (CDS) and Digital Remote Patient Monitoring (dRPM) through Virtual Care (VC) programs in Alberta to reduce length of hospital stay and readmission rates and improve long-term outcomes after AKI.

   Evidence of the effectiveness of the two digital health solutions is available from Alberta and international clinical trials. Our team previously implemented a computerized CDS intervention for AKI risk assessment and prevention and achieved improved AKI prevention and reduced AKI incidence after cardiac procedures across the province. The investigators will use a similar approach to identify high risk patients with AKI and provide recommendations to improve the quality of their care, which is well suited to the evolving digital health infrastructure in Alberta.

   Providing hospital-level care at home through Virtual Care (VC) teams has been shown to reduce mortality and readmission rates. Alberta's VC program have existed in both Edmonton and Calgary since 2018 and have reported lower readmission rates, Emergency Department (ED) visits and use of Emergency Medical Services than observed with usual care. Patients reported that the program helped them regain their independence and function. Alberta's VC programs have implemented dRPM technology, which has been further associated with fewer days in hospital and emergency department visits. Patients reported better quality of care using this technology. The framework for dRPM and complex care planning is already in place in Alberta's Virtual Care programs. The investigators intend to utilize these programs to improve transitions of care through early facilitated discharge and enhanced follow-up of patients with AKI at high risk of hospital readmission, who require frequent monitoring and more intensive care strategies during this vulnerable period of transition in care.
2. Research Question and Objectives

   * Implement and evaluate a transition of care intervention for patients with AKI.
   * Integrate digital health solutions that can achieve levels of monitoring and care in a patient's own home that are comparable to acute care, while transitioning care to the community setting.
   * Reduce the length of hospital stay and risk of hospital readmission for people with AKI.
   * Improve the long-term outcomes after hospitalization with AKI.
3. Methods

The investigators will evaluate implementation initially in a Vanguard phase to establish feasibility and acceptability of the intervention, followed by an evaluation of implementation and effectiveness of the intervention in a larger Multicenter Randomized Controlled Trial (RCT). High risk patients with AKI and a predicted risk of readmission or death ≥20% will be identified using a Best Practice Alert (BPA) in Connect Care and participants will be randomized to care with or without virtual monitoring through the VC programs. All patients will receive the same baseline interventions refined in the Vanguard phase, while the intervention arm will additionally receive VC with dRPM following discharge.

High risk patients in the intervention arm will be navigated through the transition of care pathway by a trained nurse navigator. Patients will receive dRPM kits, and biometric data will be automatically uploaded to the web-based monitoring platform and reviewed by the nurse navigator. Patients will receive regular virtual assessments via telephone or videoconferencing (via the tablet) after in-patient discharge. Blood tests will be drawn at home by community paramedics as deemed necessary by the clinical team to assess kidney function and monitor for complications of AKI. Should concerns be identified that warrant in-person assessment, paramedic care teams will be sent for assessment and/or intervention. Upon completion of the intervention patients will be assessed for readiness to move to the subacute arms of the program and return to their primary care provider. If ongoing nephrologist or other specialist care is required, the nurse navigator will ensure appropriate follow up is arranged.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* AKI identified in hospital using Kidney Disease Improving Global Outcomes (KDIGO) criteria17.
* Hospitalization > 48 hours.
* LACE (L= Length patient Stay in the hospital, A= Acuity of Admission of patient in the hospital, C= Comorbidity and E= Emergency Visit.) Score 12 or higher.
* Meets all inclusion criteria of Virtual Home Hospital programs of Calgary and Edmonton zones.

Exclusion Criteria:

* Non-Alberta residents.
* Resides outside the catchment areas for the Calgary and Edmonton Virtual Home Hospital programs.
* C1 or C2 goals of care.
* Hospitalization > 30 days.
* Will be discharged to long-term care.
* Kidney failure receiving dialysis.
* Already admitted in Virtual Home Hospital Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
the number of days alive out of hospital | Up to 45 days from the date of randomization
  the number of days alive out of hospital

SECONDARY OUTCOMES:
the time as inpatient in hospital | Up to 45 days from the date of randomization
  the time as inpatient in hospital
death | from the date of randomization up to 45 days, or date of death from any cause, whichever came first,
  death records from health administrative data.
hospital readmission | Up to 45 days from the date of randomization
  hospital readmission records from health administrative data.
Emergency Department visits | Up to 45 days from the date of randomization
  Emergency Department visit records from health administrative data.
Estimated Glomerular Filtration (eGFR) | At 90 days after the date of randomization
  eGFR
Urine Albumin Creatinine Ration (ACR) | At 90 days after the date of randomization
  ACR laboratory test
total number of physician visits | Up to 45 days from the date of randomization
  total number of physician visits
number of physician visits by specialty | Up to 45 days from the date of randomization
  primary care vs. non-primary care
Changes to medication prescription | Up to 45 days from the date of randomization
  Changes to medication prescription (including starting, stopping, or dose adjustment) of an Angiotensin-Converting Enzyme Inhibitors (ACEI)/Angiotensin receptor blockers (ARB), diuretic, SGLT2 inhibitor, or NSAID or administration of IV fluid
laboratory testing | Up to 45 days from the date of randomization
  Number of creatinine/eGFR, electrolytes, and urine protein quantification
patient experience care transition measure | At 45 days after the date of randomization
  Online Survey
Euro Qol- 5 Dimension (EQ5D) | At 45 days after the date of randomization
  Online Survey to assess quality of life mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" to "extreme problems

CONTACTS AND LOCATIONS:
Overall Officials: Matthew James, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Background] Kawamoto K, Houlihan CA, Balas EA, Lobach DF. Improving clinical practice using clinical decision support systems: a systematic review of trials to identify features critical to success. BMJ. 2005 Apr 2;330(7494):765. doi: 10.1136/bmj.38398.500764.8F. Epub 2005 Mar 14. PMID 15767266
- [Background] Roshanov PS, Fernandes N, Wilczynski JM, Hemens BJ, You JJ, Handler SM, Nieuwlaat R, Souza NM, Beyene J, Van Spall HG, Garg AX, Haynes RB. Features of effective computerised clinical decision support systems: meta-regression of 162 randomised trials. BMJ. 2013 Feb 14;346:f657. doi: 10.1136/bmj.f657. PMID 23412440
- [Background] James MT, Har BJ, Tyrrell BD, Faris PD, Tan Z, Spertus JA, Wilton SB, Ghali WA, Knudtson ML, Sajobi TT, Pannu NI, Klarenbach SW, Graham MM. Effect of Clinical Decision Support With Audit and Feedback on Prevention of Acute Kidney Injury in Patients Undergoing Coronary Angiography: A Randomized Clinical Trial. JAMA. 2022 Sep 6;328(9):839-849. doi: 10.1001/jama.2022.13382. PMID 36066520
- [Background] James MT, Har BJ, Tyrrell BD, Ma B, Faris P, Sajobi TT, Allen DW, Spertus JA, Wilton SB, Pannu N, Klarenbach SW, Graham MM. Clinical Decision Support to Reduce Contrast-Induced Kidney Injury During Cardiac Catheterization: Design of a Randomized Stepped-Wedge Trial. Can J Cardiol. 2019 Sep;35(9):1124-1133. doi: 10.1016/j.cjca.2019.06.002. Epub 2019 Jun 7. PMID 31472811
- [Background] Caplan GA, Sulaiman NS, Mangin DA, Aimonino Ricauda N, Wilson AD, Barclay L. A meta-analysis of "hospital in the home". Med J Aust. 2012 Nov 5;197(9):512-9. doi: 10.5694/mja12.10480. PMID 23121588
- [Background] Goncalves-Bradley DC, Iliffe S, Doll HA, Broad J, Gladman J, Langhorne P, Richards SH, Shepperd S. Early discharge hospital at home. Cochrane Database Syst Rev. 2017 Jun 26;6(6):CD000356. doi: 10.1002/14651858.CD000356.pub4. PMID 28651296
- [Background] Grinman, M., Kozicky, R. & Smith, M. Bringing Acute General Internal Medicine Outside of Hospital Walls. Canadian Journal of General Internal Medicine 17, 548 (2022
- [Background] Gibbons-Reid, V., Wodinski, L. & Reynolds, C. Early Adoption & Implementation of Digital Remote Patient Monitoring in Virtual Hospital Care: Evaluation Report. Health Systems Evaluation and Evidence. (2021).
- [Background] McGillion MH, Parlow J, Borges FK, Marcucci M, Jacka M, Adili A, Lalu MM, Ouellette C, Bird M, Ofori S, Roshanov PS, Patel A, Yang H, O'Leary S, Tandon V, Hamilton GM, Mrkobrada M, Conen D, Harvey V, Lounsbury J, Mian R, Bangdiwala SI, Arellano R, Scott T, Guyatt GH, Gao P, Graham M, Nenshi R, Forster AJ, Nagappa M, Levesque K, Marosi K, Chaudhry S, Haider S, Deuchar L, LeBlanc B, McCartney CJL, Schemitsch EH, Vincent J, Pettit SM, DuMerton D, Paulin AD, Simunovic M, Williams DC, Halman S, Harlock J, Meyer RM, Taylor DA, Shanthanna H, Schlachta CM, Parry N, Pichora DR, Yousuf H, Peter E, Lamy A, Petch J, Moloo H, Sehmbi H, Waggott M, Shelley J, Belley-Cote EP, Devereaux PJ; PVC-RAM-1 Investigators. Post-discharge after surgery Virtual Care with Remote Automated Monitoring-1 (PVC-RAM-1) technology versus standard care: randomised controlled trial. BMJ. 2021 Sep 30;374:n2209. doi: 10.1136/bmj.n2209. PMID 34593374